CLINICAL TRIAL: NCT01472822
Title: Efficacy and Safety of Omija Extract on Gonarthritis
Brief Title: Efficacy of Omija (Schisandra Chinensis) Extract in Subjects With Knee Osteoarthritis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Chonbuk National University Hospital (Other)
Responsible Party: Principal Investigator, Soo-Wan Chae, Clinical Trial Center for Functional Foods, Chonbuk National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: BIOYD-KA-SCHISANDRA
Record Dates: First submitted 2011-11-14; First posted 2011-11-17 (Estimated); Results first posted 2013-02-04 (Estimated); Last update posted 2013-02-04 (Estimated); Status verified 2012-12

CONDITIONS: Mild Knee Osteoarthritis
Keywords: Omija; knee osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Omija extract. (Experimental)
  Interventions: Dietary Supplement: Omija extract.
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Omija extract. — Omija extract 1.2g/day for 12weeks
  Arms: Omija extract.
Dietary Supplement: Placebo — Placebo 1.2g/day for 12weeks
  Arms: Placebo

SUMMARY:
Knee osteoarthritis (KO) is a common arthropathy and a leading cause of disability in elderly adults. Schizandra chinensis(Omija) has been known to have five predominant tastes: salty, sweet, sour, astringent, and bitter. It has also been shown to have various effects on the anti-inflammatory, cardiovascular system, gastrointestinal system, central nervous system, endocrine system, and stress protect. Therefore, this study is designed to evaluate the efficacy and safety on KO of Omija extract.

DETAILED DESCRIPTION:
In the present study, the investigators will assess the efficacy and safety of the formulation of Omija extract(1,200 mg administered twice a day) on the symptoms of knee osteoarthritis (KO) during a 12-week treatment course. In a randomized, double-blind placebo-controlled trial, subjects will be randomly assign to receive oral omija treatment group(n=30) or placebo group(n=30). The primary efficacy outcome measure will be score change in the WOMAC(Western Ontario and McMaster University Osteoarthritis Index) after 12-weeks. Secondary parameters will be included the Lysholm index score, hs-CRP, osteocalcin(OSC), and deoxypyridinoline(DPYR).

ELIGIBILITY:
Inclusion Criteria:

* Males and females 30-70 years old
* mild to Moderate KO(Knee Osteoarthritis) as indicated by WOMAC(Western Ontario and McMaster University Osteoarthritis Index) score ≥ 38
* Able to walk
* Subject agrees not to start any new therapies for OA during the course of the study
* Able to give informed consent

Exclusion Criteria:

* History of underlying inflammatory arthropathy; septic arthritis; inflammatory joint disease; gout; pseudogout; Paget's disease; joint fracture; acromegaly; fibromyalgia; Wilson's disease; ochronosis; haemochromatosis; heritable arthritic disorder or collagen gene mutations or rheumatoid arthritis
* Expectation of surgery in the next 4 months
* Recent injury in the area affected by OA of the knee, i.e. meniscal tear (past 4 months)
* Cartilage reconstruction procedure in the target knee
* Intra-articular corticosteroid injections in the target knee within the last 3 months
* Viscous injections in the target knee within the last 6 months
* Abnormal liver or kidney function tests (ALT or AST > 2 times the upper limit of normal; elevated creatinine, males>125 umol/L, females>110 umol/L)

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-03; Primary Completion 2011-06 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeong-Hwan Seo, MD, Principal Investigator — Chonbuk National University Hospital
Locations (1):
- Clinical Trial Center for Functional Foods; Chonbuk National University Hospital, Jeonju, Jeollabuk-do, South Korea

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through local advertising and doctor referrals from hospital outpatients and general practice clinics.
Pre-assignment Details: The criteria were an age from 30 to 70 years, mild to Moderate KO as indicated by WOMAC(Western Ontario and McMaster Universities Arthritis Index) score ≥ 38 subjects.
Groups:
- Omija Extract.: Omija extract.(2times/day, 4tablets/day, 1.2g/day) for 12weeks
  Omija extract.: Omija extracted with ethanol and then concentrated and dried.
- Placebo: Placebo(2times/day, 4tablets/day, 1.2g/day) for 12weeks
  Placebo : Amount and calorie of placebo are same with Omija extract..
Period: Overall Study
Arm/Group | Omija Extract. | Placebo
Started | 30 | 30
Completed | 28 | 28
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Omija | Placebo | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 30 | 60
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 52.1 (9.5) | 52.4 (9.6) | 52.2 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 28 | 55
  Male | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Changes in WOMAC (Western Ontario and McMaster University Osteoarthritis Index) Totol Score
Description: WOMAC(Western Ontario and McMaster University Osteoarthritis Index) total score (score 0-96) was measured in study visit 1(0 week) and visit 3(12 week).
  The original index consists of 24 Questions. Individual question response is assigned a score of between 0 (none) to 4 (extreme) and summed to form a score ranging from 0 (best) to 96 (worst).
Time Frame: 12 weeks
Population: per protocol analysis
Measure: Mean (Standard Deviation); unit: Score
Groups:
- Omija Extract: Oral intake Omija extract(1.2g/day) for 12weeks.
- Placebo: Oral intake placebo(1.2g/day) for 12weeks
Arm/Group | Omija Extract | Placebo
Number analyzed (Participants) | 28 | 28
Score
  Visit 1(0 week) | 56.0 (11.6) | 53.3 (11.3)
  visit 3(12 week) | 34.8 (17.2) | 31.5 (15.5)

2. Secondary Outcome: Changes in Lysholm Index Score
Description: Lysholm index score total score (score 0-100) was measured in study visit 1(0 week) and visit 3(12 week).
  The original index consists of 9 Questions(Limp, Assive devices, Up stair, Giving way, Sauat, Sit down&up, Cripitation, Swelling, Pain). Lysholm index score total score summed to form a score ranging from 0 (worst) to 100 (best).
Time Frame: 12 weeks
Population: per protocol analysis
Measure: Mean (Standard Deviation); unit: units on a scale(0-100)
Arm/Group | Omija Extract | Placebo
Number analyzed (Participants) | 28 | 28
units on a scale(0-100)
  Visit 1(0 week) | 52.6 (11.0) | 48.3 (13.1)
  Visit 3(12 week) | 54.8 (10.8) | 59.9 (15.6)

3. Secondary Outcome: Changes in Hs-CRP(High Sensitivity C-reactive Protein)
Description: hs-CRP(high sensitivity C-reactive protein) was measured in study visit 1(0 week) and visit 3(12 week).
Time Frame: 12 weeks
Population: per protocol analysis
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Omija Extract | Placebo
Number analyzed (Participants) | 28 | 28
mg/L
  Visit 1(0 week) | 0.3 (0.4) | 1.2 (4.3)
  Visit 3(12 week) | 0.5 (0.9) | 0.6 (1.1)

4. Secondary Outcome: Changes in OSC(Osteocalcin)
Description: OSC(Osteocalcin) was measured in study visit 1(0 week) and visit 3(12 week).
Time Frame: 12 weeks
Population: per protocol analysis
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Omija Extract | Placebo
Number analyzed (Participants) | 28 | 28
ng/ml
  Visit 1(0 week) | 16.5 (6.2) | 16.6 (7.0)
  Visit 3(12 week) | 16.8 (5.3) | 17.3 (7.4)

5. Secondary Outcome: Changes in DPD(Deoxypyridinoline)
Description: DPD(Deoxypyridinoline) was measured in study visit 1(0 week) and visit 3(12 week).
Time Frame: 12 weeks
Population: per protocol analysis
Measure: Mean (Standard Deviation); unit: nanoMolar DPD per milliMolar creatine
Arm/Group | Omija Extract | Placebo
Number analyzed (Participants) | 28 | 28
nanoMolar DPD per milliMolar creatine
  Visit 1(0 week) | 7.3 (2.5) | 7.2 (2.7)
  Visit 3(12 week) | 7.2 (1.9) | 7.5 (2.0)

ADVERSE EVENTS:
Description: Serious and/or other [non-serious] adverse events were not collected/assessed
Arm/Group | Omija | Placebo
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No